CLINICAL TRIAL: NCT02762227
Title: The Role of Different Imaging Methods in the Diagnosis of Gallbladder Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RenJiH
Record Dates: First submitted 2016-03-28; First posted 2016-05-04 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2019-10

CONDITIONS: Polyp of Gallbladder
Keywords: CEUS; CT; gallbladder cholesterol polyps; adenoma; gallbladder cancer
MeSH Terms: conditions — Adenoma; Gallbladder Neoplasms | interventions — Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gallbladder polyps patients (Experimental): All patients with a gallbladder polypoid lesion visited our department, diagnosed by conventional transabdominal US, were enrolled in this study.
  Of these patients, we excluded: (1) gallbladder polyp with a diameter less than 10 mm. (2) lesions highly suspected to be cancer due to visible metastasis. (3) allergy to contrast agents and cannot received CT or CEUS examination. (4) women in pregnancy or lactation.
  All patients received transabdominal US, abdominal high resolution CT and contrast-enhanced ultrasonography (CEUS) before the cholecystectomy.
  Interventions: Device: Abdominal high resolution CT; Device: Contrast-enhanced ultrasonography (CEUS); Procedure: Cholecystectomy

INTERVENTIONS:
Device: Abdominal high resolution CT — CT examinations were performed using a 64-slice CT scanner. Arterial phase scanning was triggered by bolus tracking technique after 100 to 120 mL nonionic contrast material was injected through the antecubital vein. With a delay of 60 and 140 s after the beginning of contrast medium injection, portal venous and equilibrium phase image scanning were followed.
Device: Contrast-enhanced ultrasonography (CEUS) — CEUS examinations were performed using a Philips iU 22 scanner with a 1-5 MHz（Mega Hertz, MHz）vector transducer. Traditional transabdominal ultrasound and CEUS were performed by the same investigator, one with more than 3 years experiences in CEUS. Traditional ultrasound was used initially to locate the lesion. The plane with the bottom of the lesion was selected for further examination. When multiple lesions were existed, the largest one was selected to evaluate. The target was placed in the center of the screen and was kept stable. Pulse inversion harmonic imaging with an index of 0.06 was used in CEUS examination. SonoVue, which contained sulfur hexafluoride microbubbles, was used as the contrast agent.
Procedure: Cholecystectomy — Cholecystectomy is performed by method of either laparoscopic cholecystectomy or open cholecystectomy.

SUMMARY:
This prospective cohort study is designed to investigate and to compare the diagnostic performance of contrast-enhanced ultrasonography (CEUS) and multidetector computed tomography (CT) for gallbladder cholesterol polyps, adenoma and gallbladder cancer.

DETAILED DESCRIPTION:
In this study, investigators aimed to investigate the diagnostic performance of CEUS and high resolution CT (HRCT) for the preoperative differential diagnostic accuracies of gallbladder polypoid lesions.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a gallbladder polypoid lesion visited our department, diagnosed by conventional transabdominal US.

Exclusion Criteria:

* Gallbladder polyp with a diameter less than 10 mm.
* Lesions highly suspected to be cancer due to visible metastasis.
* Allergy to contrast agents and cannot received CT or CEUS examination.
* Women in pregnancy or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pathological diagnosis of gallbladder polyps （Cholesterol / Adenoma / Others） | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: JIAN WANG, M.D., Principal Investigator — Department of Biliary-pancreatic Surgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- RenJi Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No